CLINICAL TRIAL: NCT02637804
Title: Daily Disposable Silicone Hydrogel Contact Lens, Stenfilcon A, Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JP-MKTG-201512
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Results first posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Study participants will be allocated in to 2 parallel groups: Group 1: stenfilcon A and narafilcon A, and Group 2: stenfilcon A and delefilcon A. Each participant will be randomized to wear either lens pair in a bilateral design for 1 week, and then cross over to the alternative pair.
Oversight: Data Monitoring Committee: No

ARMS (2):
- stenfilcon A vs narafilcon A (Group 1) (Active Comparator): Participants are randomized to wear either stenfilcon A lens pair or narafilcon A lens pair, bilaterally, for 1 week during the cross over study.
  Interventions: Device: stenfilcon A; Device: narafilcon A
- stenfilcon A vs delefilcon A (Group 2) (Active Comparator): Participants are randomized to wear either stenfilcon A lens pair or delefilcon A lens pair, bilaterally, for 1 week during the cross over study.
  Interventions: Device: stenfilcon A; Device: delefilcon A

INTERVENTIONS:
Device: stenfilcon A — contact lens
Device: narafilcon A — contact lens
  Arms: stenfilcon A vs narafilcon A (Group 1)
Device: delefilcon A — contact lens
  Arms: stenfilcon A vs delefilcon A (Group 2)

SUMMARY:
Clinical evaluation of stenfilcon A compared with narafilcon A and delefilcon A

This is a total 120 subject, randomized, open label, bilateral wear, two week crossover study (each lens for 1 week) evaluating the clinical performance of stenfilcon A spherical lenses compared to narafilcon A or delefilcon A spherical lenses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the clinical performance of stenfilcon A compared with narafilcon A and delefilcon A.

The study participants will be allocated to two parallel groups (Group 1 and Group 2), 60 subjects each, based on the control lenses, narafilcon A and delefilcon A spherical lenses.

Study groups:

Group 1: stenfilcon A vs. narafilcon A

Group 2: stenfilcon A vs. delefilcon A

ELIGIBILITY:
Inclusion Criteria:

- A person is eligible for inclusion in the study if he/she:

* Is over 18 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted daily disposable non-silicone hydrogel spherical contact lens wearer
* Can achieve best corrected spectacle distance visual acuity of 20/25 or better in each eye.
* Can achieve a distance visual acuity of 20/30 or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Has a CL (Contact Lens) spherical prescription between - 0.75 and - 8.00 (inclusive)
* Is willing to comply with the wear schedule.
* Is willing to comply with the visit schedule

Exclusion Criteria:

- A person will be excluded from the study if he/she:

* Is not a habitual wearer of daily disposable non-silicone hydrogel spherical contact lenses
* Has a CL prescription outside the range of the inclusion power range
* Has a spectacle cylinder ≥1.00D of cylinder in either eye.
* Has a history of not achieving comfortable CL wear (5 days per week; > 8 hours/day)
* Has contact lens best corrected distance vision worse than 20/25 in either eye
* Presence of clinically significant (grade 2-4) anterior segment abnormalities
* Presence of ocular or systemic disease or need of medications which might interfere with contact lens wear
* Slit lamp findings that would contraindicate contact lens wear
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kodama, MD, PhD, Principal Investigator — Director, Kodama Eye Clinic

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Stenfilcon A, Then Narafilcon A (Group 1); Narafilcon A, Then Stenfilcon A (Group 1): Participants are randomized to wear either stenfilcon A lens pair or narafilcon A lens pair, bilaterally, for 1 week during the cross over study.
  stenfilcon A: contact lens
  narafilcon A: contact lens
- Stenfilcon A, Then Delefilcon A (Group 2); Delefilcon A, Then Stenfilcon A (Group 2): Participants are randomized to wear either stenfilcon A lens pair or delefilcon A lens pair, bilaterally, for 1 week during the cross over study.
  stenfilcon A: contact lens
  delefilcon A: contact lens
Period: First Intervention (1 Week)
Arm/Group | Stenfilcon A, Then Narafilcon A (Group 1) | Narafilcon A, Then Stenfilcon A (Group 1) | Stenfilcon A, Then Delefilcon A (Group 2) | Delefilcon A, Then Stenfilcon A (Group 2)
Started | 27 | 28 | 25 | 26
Completed | 27 | 28 | 25 | 26
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Stenfilcon A, Then Narafilcon A (Group 1) | Narafilcon A, Then Stenfilcon A (Group 1) | Stenfilcon A, Then Delefilcon A (Group 2) | Delefilcon A, Then Stenfilcon A (Group 2)
Started | 27 | 28 | 25 | 26
Completed | 27 | 28 | 25 | 26
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Characteristics - Group 1:Stenfilcon A & Narafilcon A: Participants are randomized to wear either stenfilcon A lens pair or narafilcon A lens pair, bilaterally, for 1 week during the cross over study.
  stenfilcon A: contact lens
  narafilcon A: contact lens
- Overall Characteristics - Group 2: Stenfilcon A & Delefilcon A: Participants are randomized to wear either stenfilcon A lens pair or delefilcon A lens pair, bilaterally, for 1 week during the cross over study.
  stenfilcon A: contact lens
  delefilcon A: contact lens
- Total: Total of all reporting groups
Arm/Group | Overall Characteristics - Group 1:Stenfilcon A & Narafilcon A | Overall Characteristics - Group 2: Stenfilcon A & Delefilcon A | Total
Number analyzed (Participants) | 55 | 51 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11) | 33 (11) | 34 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 88
  Male | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  Japan | 55 | 51 | 106

OUTCOME MEASURES:

1. Primary Outcome: Pain and Foreign Body Sensation
Description: Subjective ratings of pain and foreign body sensation for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at 1 week. Grade 0-3, 0=No sensation, 1=Slightly: sometimes felt sensation without any trouble in wearing contact lenses, 2=Mild: always felt sensation without any trouble in wearing contact lenses, 3=Heavy: could not wear contact lense due to sensation
Time Frame: 1 week
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Groups:
- Stenfilcon A (Group 1); Narafilcon A (Group 1): Participants are randomized to wear either stenfilcon A lens pair or narafilcon A lens pair, bilaterally, for 1 week during the cross over study.
  stenfilcon A: contact lens
  narafilcon A: contact lens
- Stenfilcon A (Group 2); Delefilcon A (Group 2): Participants are randomized to wear either stenfilcon A lens pair or delefilcon A lens pair, bilaterally, for 1 week during the cross over study.
  stenfilcon A: contact lens
  delefilcon A: contact lens
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
eyes
  No sensation | 89 | 79 | 83 | 87
  Slight sensation | 21 | 28 | 19 | 13
  Mild sensation | 0 | 3 | 0 | 2
  Heavy sensation | 0 | 0 | 0 | 0

2. Primary Outcome: Itching Sensation on Removal
Description: Subjective ratings of itching sensation on insertion for each lens pair assessed at 1 week. Grade 0-3, 0=No sensation, 1=Slightly: sometimes felt sensation without any trouble in wearing contact lenses, 2=Mild: always felt sensation without any trouble in wearing contact lenses, 3=Heavy: could not wear contact lense due to sensation
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  No sensation | 98 | 102 | 92 | 90
  Slight sensation | 9 | 8 | 10 | 10
  Mild sensation | 3 | 0 | 0 | 0
  Heavy sensation | 0 | 0 | 0 | 2

3. Primary Outcome: Red Eye Sensation
Description: Subjective ratings of red eye sensation for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at 1 week. Grade 0-3, 0=No sensation, 1=Slightly: sometimes felt sensation without any trouble in wearing contact lenses, 2=Mild: always felt sensation without any trouble in wearing contact lenses, 3=Heavy: could not wear contact lense due to sensation
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  No sensation | 98 | 98 | 92 | 87
  Slight sensation | 12 | 10 | 8 | 15
  Mild sensation | 0 | 2 | 2 | 0
  Heavy sensation | 0 | 0 | 0 | 0

4. Primary Outcome: Dryness
Description: Subjective ratings of dryness (right after insertion, right before removal, all day long) for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at 1 week. (Scale 0-10, 0=very dry, 10=no dryness at all.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
units on a scale
  Right after insertion | 9.56 (1.14) | 9.40 (1.36) | 9.84 (0.50) | 9.76 (0.90)
  Right before removal | 7.37 (2.21) | 7.70 (2.10) | 7.61 (2.02) | 7.71 (2.45)
  All day long | 8.08 (1.89) | 8.36 (1.74) | 8.27 (1.66) | 8.40 (1.92)

5. Primary Outcome: Comfort
Description: Subjective ratings of comfort (right after insertion, right before removal, all day long) for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at 1 week. (Scale 0-10, 0=very poor comfort, 10=very good comfort).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
units on a scale
  Right after insertion | 9.22 (1.43) | 9.16 (1.52) | 9.67 (0.63) | 9.69 (0.62)
  Right before removal | 8.00 (1.85) | 8.17 (2.00) | 8.43 (2.02) | 8.29 (1.94)
  All day long | 8.49 (1.72) | 8.52 (1.76) | 8.86 (1.48) | 8.67 (1.67)

6. Primary Outcome: Vision
Description: Subjective ratings of vision (right after insertion, right before removal, all day long) for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at 1 week. (Scale 0-10, 0=very poor vision, 10=very good vision).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
units on a scale
  Right after insertion | 9.29 (1.55) | 9.32 (1.40) | 9.66 (0.81) | 9.57 (0.90)
  Right before removal | 8.46 (1.76) | 8.52 (2.08) | 8.87 (1.18) | 8.83 (1.61)
  All day long | 8.80 (1.59) | 8.81 (1.76) | 9.13 (0.94) | 9.02 (1.35)

7. Primary Outcome: Handling
Description: Subjective ratings of handling (lens insertion and lens removal) for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at 1 week. (Scale 0-10, 0=very poor handling, 10=very good handling.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
units on a scale
  Lens insertion | 9.07 (1.54) | 9.64 (0.92) | 9.27 (1.50) | 9.33 (1.33)
  Lens removal | 8.63 (1.72) | 9.32 (1.25) | 8.88 (1.75) | 7.63 (2.62)

8. Primary Outcome: Lens Preference - Stenfilcon A/Narafilcon A (Group 1)
Description: Subjective ratings of lens preference for stenfilcon A/narafilcon A assessed at 1 week. (5 possible ratings: Prefer stenfilcon A, Little Prefer stenfilcon A, No preference, little prefer narafilcon A, prefer narafilcon A).
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Prefer Stenfilcon A; Little Prefer Stenfilcon A: stenfilcon A: contact lens
- No Preference: No Preference
- Little Prefer Narafilcon A; Prefer Narafilcon A: narafilcon A: contact lens
Arm/Group | Prefer Stenfilcon A | Little Prefer Stenfilcon A | No Preference | Little Prefer Narafilcon A | Prefer Narafilcon A
Number analyzed (Participants) | 55 | 55 | 55 | 55 | 55
Participants | 15 | 12 | 5 | 10 | 13

9. Primary Outcome: Lens Preference - Stenfilcon A/Delefilcon A (Group 2)
Description: Subjective ratings of lens preference for stenfilcon A/narafilcon A assessed at 1 week. (5 possible ratings: Prefer stenfilcon A, Little Prefer stenfilcon A, No preference, little prefer delefilcon A, prefer delefilcon A).
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Little Prefer Delefilcon A; Prefer Delefilcon A: delefilcon A: contact lens
Arm/Group | Prefer Stenfilcon A | Little Prefer Stenfilcon A | No Preference | Little Prefer Delefilcon A | Prefer Delefilcon A
Number analyzed (Participants) | 51 | 51 | 51 | 51 | 51
Participants | 14 | 8 | 3 | 9 | 17

10. Secondary Outcome: Lens Fit - Horizontal Centration
Description: Lens fit evaluation of horizontal centration for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at baseline. (Temporal, Little temporal, Centered, Little nasal, Nasal)
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Temporal | 0 | 0 | 0 | 0
  Little Temporal | 1 | 6 | 0 | 2
  Central | 109 | 104 | 102 | 100
  Little Nasal | 0 | 0 | 0 | 0
  Nasal | 0 | 0 | 0 | 0

11. Secondary Outcome: Lens Fit - Horizontal Centration
Description: Lens fit evaluation of horizontal centration for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A assessed at 1 week. (Temporal, Little temporal, Centered, Little nasal, Nasal)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Temporal | 0 | 0 | 0 | 0
  Little Temporal | 0 | 8 | 0 | 1
  Central | 110 | 102 | 102 | 100
  Little Nasal | 0 | 0 | 0 | 1
  Nasal | 0 | 0 | 0 | 0

12. Secondary Outcome: Lens Fit - Vertical Centration
Description: Lens fit evaluation of vertical centration for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at baseline. (Upper, Little upper, Centered, Little lower, Lower)
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Upper | 0 | 0 | 0 | 0
  Little Upper | 2 | 16 | 0 | 4
  Central | 104 | 86 | 100 | 96
  Little Lower | 4 | 8 | 2 | 2
  Lower | 0 | 0 | 0 | 0

13. Secondary Outcome: Lens Fit - Vertical Centration
Description: Lens fit evaluation of vertical centration for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Upper, Little upper, Centered, Little lower, Lower)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Upper | 0 | 0 | 0 | 0
  Little Upper | 0 | 7 | 0 | 4
  Central | 107 | 90 | 102 | 98
  Little Lower | 3 | 13 | 0 | 0
  Lower | 0 | 0 | 0 | 0

14. Secondary Outcome: Lens Fit - Post-blink Movement
Description: Lens fit evaluation of post-blink movement for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at baseline. (Tight, Little tight, Optimal, Little loose, Loose)
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Tight | 0 | 0 | 0 | 0
  Little Tight | 0 | 6 | 2 | 4
  Optimum | 104 | 94 | 96 | 97
  Little Loose | 6 | 10 | 4 | 1
  Loose | 0 | 0 | 0 | 0

15. Secondary Outcome: Lens Fit - Post-blink Movement
Description: Lens fit evaluation of post-blink movement for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Tight, Little tight, Optimal, Little loose, Loose)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Tight | 0 | 2 | 0 | 0
  Little Tight | 0 | 10 | 1 | 5
  Optimum | 107 | 92 | 97 | 97
  Little Loose | 3 | 5 | 4 | 0
  Loose | 0 | 1 | 0 | 0

16. Secondary Outcome: Lens Fit Overall
Description: Lens fit evaluation overall for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at baseline. (Optimum, Good, Acceptable, Not acceptable (cannot wear))
Time Frame: Baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Optimum | 100 | 81 | 96 | 90
  Good | 10 | 26 | 4 | 12
  Acceptable | 0 | 3 | 2 | 0
  Not Acceptable | 0 | 0 | 0 | 0

17. Secondary Outcome: Lens Fit Overall
Description: Lens fit evaluation overall for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Optimum, Good, Acceptable, Not acceptable (cannot wear))
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Optimum | 102 | 75 | 98 | 95
  Good | 8 | 30 | 2 | 7
  Acceptable | 0 | 3 | 2 | 0
  Not Acceptable | 0 | 2 | 0 | 0

18. Secondary Outcome: Conjunctival Redness
Description: Conjunctival redness for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Grading scale 0-4, 0.5 steps 0=Normal, 1=Trace 2=MIld, 3=Moderate 4=Severe)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Normal | 104 | 99 | 100 | 100
  Trace | 6 | 11 | 2 | 2
  Mild | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

19. Secondary Outcome: Limbal Redness
Description: Limbal redness for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Grading scale 0-4, 0.5 steps 0=Normal, 1=Trace 2=MIld, 3=Moderate 4=Severe)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Normal | 110 | 106 | 102 | 99
  Trace | 0 | 4 | 0 | 3
  Mild | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

20. Secondary Outcome: Corneal Staining
Description: Corneal staining for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Grading scale 0-4, 0.5 steps 0=Normal, 1=Trace 2=MIld, 3=Moderate 4=Severe)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Normal | 83 | 69 | 71 | 70
  Trace | 25 | 39 | 31 | 29
  Mild | 2 | 2 | 0 | 3
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

21. Secondary Outcome: Corneal Neovascularization
Description: Corneal neovascularization for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Grading scale 0-4, 0.5 steps 0=Normal, 1=Trace 2=MIld, 3=Moderate 4=Severe)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Normal | 108 | 108 | 102 | 102
  Trace | 2 | 2 | 0 | 0
  Mild | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

22. Secondary Outcome: Conjunctival Staining
Description: Conjunctival staining for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Grading scale 0-4, 0.5 steps 0=Normal, 1=Trace 2=MIld, 3=Moderate 4=Severe)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Normal | 75 | 67 | 76 | 80
  Trace | 28 | 29 | 22 | 16
  Mild | 7 | 14 | 4 | 6
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

23. Secondary Outcome: Corneal Oedema
Description: Corneal oedema for for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Grading scale 0-4, 0.5 steps 0=Normal, 1=Trace 2=MIld, 3=Moderate 4=Severe)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Normal | 110 | 110 | 102 | 102
  Trace | 0 | 0 | 0 | 0
  Mild | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

24. Secondary Outcome: Papillary Conjunctivitis
Description: Papillary conjunctivitis for stenfilcon A/narafilcon A and stenfilcon A/delefilcon A is assessed at 1 week. (Grading scale 0-4, 0.5 steps 0=Normal, 1=Trace 2=MIld, 3=Moderate 4=Severe)
Time Frame: 1 week
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group 1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Number analyzed (Participants) | 55 | 55 | 51 | 51
Number analyzed (Eyes) | 110 | 110 | 102 | 102
Eyes
  Normal | 110 | 110 | 102 | 102
  Trace | 0 | 0 | 0 | 0
  Mild | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Stenfilcon A (Group 1); Narafilcon A (Group1): Participants randomized to wear either stenfilcon A lens pair or narafilcon A lens pair, bilaterally, for 1 week then cross over.
- Stenfilcon A (Group 2); Delefilcon A (Group 2): Participants randomized to wear either stenfilcon A lens pair or delefilcon A lens pair, bilaterally, for 1 week then cross over.
Arm/Group | Stenfilcon A (Group 1) | Narafilcon A (Group1) | Stenfilcon A (Group 2) | Delefilcon A (Group 2)
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other